CLINICAL TRIAL: NCT04430413
Title: Assessment of the Effect of Platelet Rich Plasma on the Healing of Operated Sacrococcygeal Pilonidal Sinus by Open Method
Brief Title: Effect of Platelet Rich Plasma on Healing of Operated Pilonidal Sinus by Open Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Gohar, Assistant Lecturer of General Surgery, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP injection in operated PNS
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Pilonidal Disease of Natal Cleft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): 50 Participants who underwent a total excision of the pilonidal sinus and the wound remained open for secondary healing.
- Group B (Active Comparator): 50 Participants who underwent the same operation with secondary healing intention but on postoperative days 4 and 12 the platelet rich plasma was injected to the surgical wound.
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — Autologous PRP obtained via double centrifugation process of the participant's blood sample. PRP was prepared by the double Spain strategy.
  Arms: Group B

SUMMARY:
The aim of the study is to assess the healing promotion effect of platelet rich plasma in patient being operated for sacrococcygeal pilonidal sinus disease by open excision

DETAILED DESCRIPTION:
Sacrococcygeal Pilonidal disease is an infection of the skin and subcutaneous tissue at or near the upper part of the natal cleft of the buttocks. Pilonidal cavities are not true cysts and lack a fully epithelialized lining; however, the sinus tracts may be epithelialized.

Pilonidal sinus disease (PNS) has an incidence of approximately 26 per 100,000 population with a male predominance of 2:1 and the mean age of those affected is from 19 to 30 years of age. It occurs rarely after the age of 45 and children.

Pilonidal sinus disease is characterized by natal cleft suppuration due to hair follicle infection. The disease results from chronic infection of hair follicles and subsequent formation of a subcutaneous abscess because of persistent folliculitis. Hair then enters the abscess cavity and provokes a foreign body tissue reaction; chronic suppuration and discharge through a midline sinus follow.

Some individuals are asymptomatic with midline pits in the sacrococcygeal area, Symptomatic Pilonidal sinus results in chronic discharging wounds that cause pain and impact upon quality of life and social function. These sinuses may become infected and present as acute abscesses. Management of these abscesses is uncontroversial and revolves around incision and drainage, however, the mode of surgical management of the chronic discharging sinus is variable, contentious, and problematic.

The Principles of Surgical strategies require eradication of the sinus tract, complete healing of the overlying skin, and prevention of recurrence. Many methods are available for surgical management of PNS which is treated by wide excision. After excision, the wound may be left open to heal with granulation tissue, or may be immediate closed with a midline closure or by using a flap (Z-plasty, karydakis, Bascom or Rhomboid flaps). However, there is not yet a consensus on the optimal treatment.

Excision and healing by granulation is still preferred due to the low recurrence rate of (3.4%) compering with other methods (20.6%) for midline closure and (10.3%) for off-midline closure but the healing time is lengthy and requires a prolonged time of daily dressing with a risk of infection and delayed wound healing. Therefore, the search for a treatment with minimal pain, accelerated healing time and a short span of time for returning to the normal daily activities is vastly pursued.

A recent method to promote the wound-healing process is the local administration of an autologous platelet concentrate suspended in plasma named as platelet rich plasma (PRP) which contains growth factors. Concentrated growth factors have been reported to accelerate wound healing by 30-40% giving a satisfactory outcome in the treatment of chronic skin and soft tissue lesions, maxillofacial and plastic surgeries by presenting these high amounts of growth factors and chemokines.

When platelets become activated, Seven fundamental protein growth factors that are actively secreted by platelet initiate all wound healing process, including platelet derived growth factor (PDGF), epidermal growth factor (EGF), transforming growth factor (TGF), vascular endothelial growth factor (VEGF), Fibroblast growth factor (FGF), connective tissue growth factor (CTGF) & insulin like growth factor (ILGF 1) all participate in the acceleration of wound-healing process.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age >18 years and <45 years.
2. All patient who underwent sacrococcygeal pilonidal sinus operation (Open method).

Exclusion Criteria:

1. Pilonidal abscess.
2. Diabetic patient.
3. HGB < 10 g/dl.
4. Platelet count < 105/ul.
5. Anticoagulant treatment.
6. Wound cavity >35cc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the wound capacity | One Year
  Evaluation of Wound volume on postoperative days till complete healing of the wound in each group and compare rate of healing in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El Sheikh University Hospital, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

REFERENCES:
- [Background] Acarturk TO, Parsak CK, Sakman G, Demircan O. Superior gluteal artery perforator flap in the reconstruction of pilonidal sinus. J Plast Reconstr Aesthet Surg. 2010 Jan;63(1):133-9. doi: 10.1016/j.bjps.2008.07.017. Epub 2008 Nov 14. PMID 19010110
- [Background] Al-Jaberi TM. Excision and simple primary closure of chronic pilonidal sinus. Eur J Surg. 2001 Feb;167(2):133-5. doi: 10.1080/110241501750070600. PMID 11266254
- [Background] McCallum I, King PM, Bruce J. Healing by primary versus secondary intention after surgical treatment for pilonidal sinus. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006213. doi: 10.1002/14651858.CD006213.pub2. PMID 17943897
- [Background] Anderson JH, Yip CO, Nagabhushan JS, Connelly SJ. Day-case Karydakis flap for pilonidal sinus. Dis Colon Rectum. 2008 Jan;51(1):134-8. doi: 10.1007/s10350-007-9150-y. Epub 2008 Jan 12. PMID 18193323
- [Background] Aksahin E, Dogruyol D, Yuksel HY, Hapa O, Dogan O, Celebi L, Bicimoglu A. The comparison of the effect of corticosteroids and platelet-rich plasma (PRP) for the treatment of plantar fasciitis. Arch Orthop Trauma Surg. 2012 Jun;132(6):781-5. doi: 10.1007/s00402-012-1488-5. Epub 2012 Mar 8. PMID 22399039
- [Derived] Gohar MM, Ali RF, Ismail KA, Ismail TA, Nosair NA. Assessment of the effect of platelet rich plasma on the healing of operated sacrococcygeal pilonidal sinus by lay-open technique: a randomized clinical trial. BMC Surg. 2020 Sep 22;20(1):212. doi: 10.1186/s12893-020-00865-x. PMID 32962673